CLINICAL TRIAL: NCT02833714
Title: Characterization of Teriflunomide's Therapeutic Mechanisms of Action in Patients With Relapsing Remitting Multiple Sclerosis.
Brief Title: Teriflunomide's Therapeutic Mechanisms of Action in Patients With Relapsing Remitting Multiple Sclerosis.
Status: Terminated | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-2877
Record Dates: First submitted 2016-06-21; First posted 2016-07-14 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: RELAPSING REMITTING MULTIPLE SCLEROSIS
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this research is to characterize the effect of teriflunomide on the activation of B-cells, as well as its capacity to modify B-cell cytokine secretion. The in-vitro identified effects of teriflunomide on the expression of B-cell activation markers, costimulatory and antigen presenting molecules, as well as on cytokine secretion, will then be confirmed in a cohort of Relapsing Remitting Multiple Sclerosis (RRMS) patients treated with this medication.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of RRMS according to McDonald's diagnostic criteria,
* age 18-55,
* an extended disability status score (EDSS) of 1.5-5.5.

Exclusion Criteria:

- Previous treatment with DMT.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Neurology/MS clinic: patients with Relapsing Remitting MS "Treatment naïve Relapsing Remitting MS patients will be recruited to provide samples for the in vitro tests. In addition, Relapsing Remitting MS patients who are already receiving treatment with teriflunomide as a part of their routine care will be recruited to obtain blood samples for the in vivo testing."
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
Percent Inhibition of activated/memory B-cells derived from RRMS patients. | 1 year

SECONDARY OUTCOMES:
Change in Cytokine Secretion Profile of T-cells stimulated by teriflunomide treatment | 1 year
Measure the effect of oral teriflunomide on the cytokine secretion as measured in the ex-vivo obtained longitudinal samples from the treated patients. | 1 year
Measure the effect of oral teriflunomide on the B cell activation as measured in the ex-vivo obtained longitudinal samples from the treated patients. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Silva MarkovicPlese, MD, Principal Investigator — Universtiy of North Carolina at Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] O'Connor P, Wolinsky JS, Confavreux C, Comi G, Kappos L, Olsson TP, Benzerdjeb H, Truffinet P, Wang L, Miller A, Freedman MS; TEMSO Trial Group. Randomized trial of oral teriflunomide for relapsing multiple sclerosis. N Engl J Med. 2011 Oct 6;365(14):1293-303. doi: 10.1056/NEJMoa1014656. PMID 21991951
- [Result] Freedman MS, Wolinsky JS, Wamil B, Confavreux C, Comi G, Kappos L, Olsson TP, Miller A, Benzerdjeb H, Li H, Simonson C, O'Connor PW; Teriflunomide Multiple Sclerosis Trial Group and the MRI Analysis Center. Teriflunomide added to interferon-beta in relapsing multiple sclerosis: a randomized phase II trial. Neurology. 2012 Jun 5;78(23):1877-85. doi: 10.1212/WNL.0b013e318258f7d4. Epub 2012 May 23. PMID 22622860
- [Result] Fox RI. Mechanism of action of leflunomide in rheumatoid arthritis. J Rheumatol Suppl. 1998 Jul;53:20-6. PMID 9666414
- [Result] Li L, Liu J, Delohery T, Zhang D, Arendt C, Jones C. The effects of teriflunomide on lymphocyte subpopulations in human peripheral blood mononuclear cells in vitro. J Neuroimmunol. 2013 Dec 15;265(1-2):82-90. doi: 10.1016/j.jneuroim.2013.10.003. Epub 2013 Oct 12. PMID 24182769
- [Result] Claussen MC, Korn T. Immune mechanisms of new therapeutic strategies in MS: teriflunomide. Clin Immunol. 2012 Jan;142(1):49-56. doi: 10.1016/j.clim.2011.02.011. Epub 2011 Mar 1. PMID 21367665
- [Result] Manna SK, Aggarwal BB. Immunosuppressive leflunomide metabolite (A77 1726) blocks TNF-dependent nuclear factor-kappa B activation and gene expression. J Immunol. 1999 Feb 15;162(4):2095-102. PMID 9973483
- [Result] Prineas JW, Wright RG. Macrophages, lymphocytes, and plasma cells in the perivascular compartment in chronic multiple sclerosis. Lab Invest. 1978 Apr;38(4):409-21. PMID 205724
- [Result] Hauser SL, Waubant E, Arnold DL, Vollmer T, Antel J, Fox RJ, Bar-Or A, Panzara M, Sarkar N, Agarwal S, Langer-Gould A, Smith CH; HERMES Trial Group. B-cell depletion with rituximab in relapsing-remitting multiple sclerosis. N Engl J Med. 2008 Feb 14;358(7):676-88. doi: 10.1056/NEJMoa0706383. PMID 18272891
- [Result] Bar-Or A, Fawaz L, Fan B, Darlington PJ, Rieger A, Ghorayeb C, Calabresi PA, Waubant E, Hauser SL, Zhang J, Smith CH. Abnormal B-cell cytokine responses a trigger of T-cell-mediated disease in MS? Ann Neurol. 2010 Apr;67(4):452-61. doi: 10.1002/ana.21939. PMID 20437580
- [Result] Kim SH, Huh SY, Lee SJ, Joung A, Kim HJ. A 5-year follow-up of rituximab treatment in patients with neuromyelitis optica spectrum disorder. JAMA Neurol. 2013 Sep 1;70(9):1110-7. doi: 10.1001/jamaneurol.2013.3071. PMID 23897062
- [Result] Serreze DV, Fleming SA, Chapman HD, Richard SD, Leiter EH, Tisch RM. B lymphocytes are critical antigen-presenting cells for the initiation of T cell-mediated autoimmune diabetes in nonobese diabetic mice. J Immunol. 1998 Oct 15;161(8):3912-8. PMID 9780157
- [Result] Yan J, Harvey BP, Gee RJ, Shlomchik MJ, Mamula MJ. B cells drive early T cell autoimmunity in vivo prior to dendritic cell-mediated autoantigen presentation. J Immunol. 2006 Oct 1;177(7):4481-7. doi: 10.4049/jimmunol.177.7.4481. PMID 16982884
- [Result] Zhong X, Gao W, Degauque N, Bai C, Lu Y, Kenny J, Oukka M, Strom TB, Rothstein TL. Reciprocal generation of Th1/Th17 and T(reg) cells by B1 and B2 B cells. Eur J Immunol. 2007 Sep;37(9):2400-4. doi: 10.1002/eji.200737296. PMID 17683116
- [Result] Sellam J, Rouanet S, Hendel-Chavez H, Abbed K, Sibilia J, Tebib J, Le Loet X, Combe B, Dougados M, Mariette X, Taoufik Y. Blood memory B cells are disturbed and predict the response to rituximab in patients with rheumatoid arthritis. Arthritis Rheum. 2011 Dec;63(12):3692-701. doi: 10.1002/art.30599. PMID 22127692
- [Result] Ramgolam VS, Sha Y, Marcus KL, Choudhary N, Troiani L, Chopra M, Markovic-Plese S. B cells as a therapeutic target for IFN-beta in relapsing-remitting multiple sclerosis. J Immunol. 2011 Apr 1;186(7):4518-26. doi: 10.4049/jimmunol.1000271. Epub 2011 Mar 2. PMID 21368231
- [Result] Zhang X, Tao Y, Troiani L, Markovic-Plese S. Simvastatin inhibits IFN regulatory factor 4 expression and Th17 cell differentiation in CD4+ T cells derived from patients with multiple sclerosis. J Immunol. 2011 Sep 15;187(6):3431-7. doi: 10.4049/jimmunol.1100580. Epub 2011 Aug 19. PMID 21856936
- [Result] Dimitrova P, Skapenko A, Herrmann ML, Schleyerbach R, Kalden JR, Schulze-Koops H. Restriction of de novo pyrimidine biosynthesis inhibits Th1 cell activation and promotes Th2 cell differentiation. J Immunol. 2002 Sep 15;169(6):3392-9. doi: 10.4049/jimmunol.169.6.3392. PMID 12218161
- [Result] Fillatreau S, Sweenie CH, McGeachy MJ, Gray D, Anderton SM. B cells regulate autoimmunity by provision of IL-10. Nat Immunol. 2002 Oct;3(10):944-50. doi: 10.1038/ni833. Epub 2002 Sep 3. PMID 12244307
- [Result] Zhang X, Tao Y, Chopra M, Ahn M, Marcus KL, Choudhary N, Zhu H, Markovic-Plese S. Differential reconstitution of T cell subsets following immunodepleting treatment with alemtuzumab (anti-CD52 monoclonal antibody) in patients with relapsing-remitting multiple sclerosis. J Immunol. 2013 Dec 15;191(12):5867-74. doi: 10.4049/jimmunol.1301926. Epub 2013 Nov 6. PMID 24198283
- [Result] Hirotani M, Niino M, Fukazawa T, Kikuchi S, Yabe I, Hamada S, Tajima Y, Sasaki H. Decreased IL-10 production mediated by Toll-like receptor 9 in B cells in multiple sclerosis. J Neuroimmunol. 2010 Apr 15;221(1-2):95-100. doi: 10.1016/j.jneuroim.2010.02.012. Epub 2010 Mar 15. PMID 20227772